CLINICAL TRIAL: NCT06169501
Title: Assessing a Mobile App-based Mindfulness Training to Improve Mental Health of Caregivers of Children With Autism Spectrum Disorder in Rural Areas
Brief Title: Mindfulness Intervention for Caregivers of Autism in Rural Environments
Acronym: MIND-CARE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was terminated, seeing new funding.
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Kahsi A. Pedersen, Principal Investigator, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2085966
Record Dates: First submitted 2023-11-13; First posted 2023-12-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Stress; Anxiety
Keywords: caregivers; autism; anxiety; stress; mindfulness; intervention; mobile app-based
MeSH Terms: conditions — Anxiety Disorders; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: This study employs a single-group assignment where participants are exposed to a mindfulness intervention for caregivers of children with autism spectrum disorders living in rural areas of Maine. The primary aim is to assess the intervention's impact on reducing caregiver stress and anxiety levels. Participants complete daily mindfulness lessons and report anxiety for up to 60 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All study participants will receive the app-based mindfulness intervention.
  Interventions: Behavioral: App-based Mindfulness Intervention

INTERVENTIONS:
Behavioral: App-based Mindfulness Intervention — Participants in the trial will engage in a 30-day app-based mindfulness program called Unwinding Anxiety that they can complete over a maximum of 60 days. During this time, they will practice short daily mindfulness lessons and respond to a set of brief questions regarding their anxiety levels. Ultimately, we want to assess whether this intervention helps these caregivers feel less stressed and anxious.

SUMMARY:
The purpose of this clinical trial is to investigate the effectiveness of a mobile app-based mindfulness program in improving the mental well-being of caregivers with a child diagnosed with autism spectrum disorder (ASD) who live in rural areas of Maine. The primary question the investigators aim to answer is whether this mindfulness intervention can reduce stress and anxiety in these rural caregivers of children with ASD. Participants in the trial will engage in a 30-day mindfulness program that they can complete over a maximum of 60 days. During this time, they will practice short daily mindfulness lessons and respond to a set of brief questions regarding their anxiety levels. Ultimately, the investigators want to assess whether this intervention helps these caregivers feel less stressed and anxious.

DETAILED DESCRIPTION:
Caregivers of children with autism spectrum disorder (ASD) often experience heightened stress, anxiety, and social isolation, leading to a reduced quality of life when compared to the general population and caregivers of children with other chronic health conditions. Rural caregivers of children with ASD face additional challenges due to limited access to diagnostic and treatment services, which result in delayed ASD diagnoses and increased emergency department utilization. These families are at an elevated risk of adverse outcomes linked to both the challenges of rural living and the responsibilities of caring for a child with ASD. Therefore, it is imperative to identify scalable and accessible mental health resources that effectively alleviate the stress and anxiety experienced by these caregivers living in remote regions.

This study aims to bridge the research gap by offering an innovative mobile-app based mindfulness-training program designed to reduce stress and anxiety. In this interventional pilot study, participants in the trial will engage in a 30-day mindfulness program that they can complete over a maximum of 60 days. During this time, they will practice short daily mindfulness lessons and respond to a set of brief questions regarding their anxiety levels. The study will also collect data at baseline, midpoint, endpoint, and 1-year follow-up to assess adherence, satisfaction, and changes in stress and anxiety over time. Stakeholder involvement has been essential in shaping the study design, ensuring its relevance, and developing pathways for future studies.

The study targets rural caregivers of children with ASD living in Maine, aiming to include a total of 40 caregivers (20 cohabitating romantic couples). By integrating both parents into the intervention framework, this study seeks to harness their unique insights, enhance intervention participation, and provide a more comprehensive approach to addressing the complex mental health challenges in this population. This holistic approach, integrating the experiences and perspectives of both parents, strives to improve caregivers' well-being while also enhancing the care they provide for their children.

ELIGIBILITY:
Inclusion Criteria:

1. The caregiver must be 18 years of age or older.
2. The caregiver must have a zip code classified as rural according to the Rural-Urban Commuting Area codes (RUCA) in the state of Maine.
3. The caregiver is currently living with a romantic partner (caregiver 2) who is also willing to participate in the study.
4. The caregiver's romantic partner (caregiver 2) must be 18 years of age or older.
5. The caregiver is defined as an adult, whether biological or non-biological parent/guardian, who currently resides with and provides care for a child with Autism Spectrum Disorder (ASD).
6. The caregiver must be able to speak and read English, regardless of whether English is their first language.
7. The caregiver must have the capacity to comprehend and sign an informed consent form.
8. The caregiver must be a legally authorized representative and cannot be a guardian or foster parent under the Department of Health and Human Services (DHHS).
9. The caregiver must affirm that their child has received a clinical diagnosis of ASD.
10. Both the caregiver and the child must reside at an address classified as rural according to the Rural-Urban Commuting Area codes (RUCA) in the state of Maine (identified by zip code).
11. The caregiver must possess a smartphone and have access to the internet.
12. The caregiver must agree to participate in online assessments, as well as the 30-day mindfulness intervention using the Unwinding Anxiety (UA) mobile app.

Exclusion Criteria:

1. Any medical condition or impairment that would hinder the participant's ability to engage in a study that involves daily visual and auditory tasks, as well as comprehension and adherence to the study protocol. Examples of such impairments include deafness, blindness, impaired decision making capacity and impaired intellectual functioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
stress | admission, daily from study admission up to 60-days, completion of mindfulness training (anytime between days 30-60, this will vary by participant), 1-year follow-up
  Parental Stress Scale (PSS). The PSS will be used to assess levels of stress experienced by caregivers with a child with autism as well as both positive and negative aspects of parenting. The PSS is a self-reported 18-item, 5-point Likert scale with responses ranging from 1 ("strongly disagree") to 5 ("strongly agree"). The total possible score ranges from 18 to 90, after summing all items; with higher scores reflecting higher caregiver stress.
anxiety | admission, daily from study admission up to 60-days, completion of mindfulness training (anytime between days 30-60, this will vary by participant), 1-year follow-up
  Generalized Anxiety Disorder-7 Scale (GAD-7). The GAD-7 is a self-reported measure that consists of seven items measuring worry and anxiety. Each item is scored on a four-point Likert scale with responses ranging from 0 ("not at all") to 3 ("extremely"). The total possible scores range from 0 to 21, after summing all items; with higher scores reflecting greater anxiety severity.

SECONDARY OUTCOMES:
intervention adherence | daily from study admission up to 60-days
  Adherence to the Unwinding Anxiety intervention will be measured by calculating the proportion of mindfulness training completed out of the 30 possible modules.
intervention satisfaction | study midpoint (anytime between days 15-30, this will vary by participant) and completion of mindfulness training (anytime between days 30-60, this will vary by participant)
  Abbreviated Acceptability Rating Profile (AARP). The AARP will be used to assess satisfaction of the Unwinding Anxiety mobile application intervention. The AARP is a self-reported 8-item, 6-point Likert scale with responses ranging from 1("strongly agree") to 6 ("strongly agree"). The total possible scores range from 8 to 48, after summing all items; with higher scores reflecting higher intervention satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kahsi A Pedersen, PhD, Principal Investigator — MaineHealth
Locations (1):
- Glickman Lauder Center of Excellence, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
Our Individual Participant Data (IPD) sharing plan promotes responsible data sharing, prioritizing participant privacy and consent. It covers de-identified demographic, behavioral, and daily experience data from a 60-day mindfulness study. Data access requires formal agreements with qualified researchers, ensuring privacy and responsible usage. Collaboration and scientific contribution are encouraged, with data security measures including encryption and REDCap usage. The plan adheres to high ethical and privacy standards, striking a balance between research advancement and participant protection. It underscores our commitment to ethical data handling, fostering scientific progress while respecting participant privacy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. End date 3-5 years.
Access Criteria: Access and Qualifications: Access to de-identified data will be granted exclusively to qualified researchers who enter into formal data sharing agreements. This approach serves to safeguard participant privacy and consent, limiting access to trusted individuals dedicated to responsible data utilization.